CLINICAL TRIAL: NCT07355868
Title: An Exploratory Clinical Study on the Intravenous Infusion of REGEND007 (Generic Airway Basal Layer Stem Cells) for Treatment of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Treatment of Chronic Obstructive Pulmonary Disease (COPD) by REGEND007 Cell Therapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REGEND007-COPD-251
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REGEND007 Cell Therapy (Experimental)
  Interventions: Biological: REGEND007

INTERVENTIONS:
Biological: REGEND007 — This study's intravenous infusion dose escalation protocol is based on a 3+3 dose escalation design, with a total of 4 dose groups. Each group included 3 subjects, and the dose is gradually increased until the maximum tolerated dose (MTD) or the maximum administered dose (MAD) is reached.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death worldwide with the characterization of obstructed airflow. In a large number of patients, diffusion function is impaired along with the progression of disease. REGEND007 cell therapy, comprised of airway basal cells with ability to regenerate lung tissue, is promising to COPD treatment. A prospective, single-arm, dose-escalation exploratory clinical study to evaluate the safety, tolerability and preliminary efficacy of different doses of REGEND007 cell therapy administered by intravenous infusion in the treatment of COPD, and to recommend appropriate treatment doses for subsequent clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Gender is not restricted; when signing the informed consent form, the age should be between 40 and 80 years old (inclusive of the boundary values);
* Diagnosed with COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) in 2025;
* During the screening process, the six-minute walk test should be ≥ 150 meters and < 600 meters;
* Voluntarily sign the informed consent form, be able to cooperate with the completion of the research-related procedures and examinations, and be able to describe or record the changes in the condition in a relatively complete manner.

Exclusion Criteria:

* Female subjects who are pregnant, breastfeeding, or planning to become pregnant within one year after using this product; or male subjects whose spouses are planning to become pregnant.
* Subjects evaluated by the investigator at the time of screening have a survival period of less than one year.
* Subjects with a current or past history of malignant tumors (excluding non-melanoma skin cancer, cervical cancer in situ, bladder cancer, thyroid cancer, and breast cancer, etc., which have a disease-free survival of more than five years and are judged by the investigator to have a relatively weak invasiveness) at the time of screening.
* Subjects diagnosed with pneumonia (including bacterial, fungal, or viral pneumonia) within 4 weeks before screening.
* Subjects who have experienced more than 4 episodes of moderate to severe acute exacerbation of COPD and required hospitalization within 1 year before screening.
* Subjects who have one or more results of pathogen or serological tests (nucleic acid, antigen, virus culture, specific IgG antibody levels) reporting novel coronavirus infection, or suspected novel coronavirus infection (manifesting symptoms such as fever, headache, fatigue, joint pain, runny nose, sore throat, and persistent cough, and the disease course is consistent with the prevalent strain) within 4 weeks before screening.
* Subjects with a history of invasive or non-invasive mechanical ventilation at the time of screening.
* Subjects evaluated by the investigator at the time of screening have active pulmonary tuberculosis, poorly controlled bronchial asthma, acute pulmonary embolism, severe pulmonary hypertension [cardiac ultrasound examination > 70 mmHg], etc.
* Subjects with severe non-pulmonary systemic diseases within 6 months before screening and evaluated by the investigator as not suitable to participate in this study, such as diabetic ketoacidosis or hyperosmolar coma, acute myocardial infarction, unstable angina pectoris, NYHA heart failure grade III/IV, stroke, liver cirrhosis with severe liver dysfunction, severe renal insufficiency, etc.
* Subjects with severe anemia, or controlled poorly granulocytopenia or thrombocytopenia at the time of screening.
* Subjects with a history of suicidal risk, psychiatric history or epilepsy history at the time of screening.
* Subjects with severe malnutrition at the time of screening.
* Subjects with 12-lead electrocardiogram showing severe arrhythmias (such as ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, atrial flutter, etc.) or abnormal conduct at II degree and above of the heart.
* Subjects who have participated in other clinical trials with intervention measures or received other biological agent treatment within 4 weeks before screening.
* Researchers, collaborating researchers, research coordinators, researchers participating in the study, or employees of the research center or their family members of the aforementioned personnel.
* Subjects considered by the investigator to be unsuitable for participation in the trial (increasing the risk of the subjects or interfering with the clinical trial).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of drug-related adverse events (AEs) | Within 12 weeks after administration
  All adverse medical events that occur from the time the subject signs the informed consent form. These can manifest as symptoms, signs, diseases, or abnormal laboratory test results, but they do not necessarily have a causal relationship with the investigational drug

SECONDARY OUTCOMES:
The time of the first occurrence of acute exacerbation of COPD (AECOPD) after administration | Within 12 weeks after the last administration
  The time of the first occurrence of acute exacerbation of COPD (AECOPD) after administration is an important indicator for assessing the severity and prognosis of the disease.
The changes in the annual incidence of AECOPD after administration compared to before administration | 12 weeks after administration
  The changes in the annual incidence of AECOPD after administration compared to before administration is an important indicator for assessing the severity and prognosis of the disease.
The change in the forced vital capacity (FVC) actual-to-predicted ratio compared to baseline | 24 hours after administration, 4 and 12 weeks after the last administration
  FVC is the full amount of air that can beexhaled with effort in a complete breath
The changes in forced expiratory volume in one second (FEV1) actual-to-predicted ratio compared to baseline | 24 hours after administration, 4 and 12 weeks after the last administration.
  FEV1 is the volume of breath exhaled with effort in one second.
The changes in the carbon monoxide diffusion capacity (DLCO) actual-to-predicted ratio compared to baseline | 24 hours after administration, 4 and 12 weeks after the last administration.
  DLCO is a measure of the conductance of CO across the alveolar-capillary membrane and its binding with hemoglobin.
Ratio of DLCO to lung volume (DLCO/VA)) | 24 hours after administration, 4 and 12 weeks after the last administration.
  DLCO/VA is also known as the diffusion constant, since the diffusion amount is affected by the alveolar ventilation volume, a decrease in alveolar ventilation volume can lead to a reduction in DLCO. Therefore, this value is often used for correction to eliminate the influence of lung volume on the diffusion amount.
The changes in the six-minute walk test (6MWT) compared to baseline | 24 hours after administration, 4 and 12 weeks after the last administration.
  6MWT is one of the commonly used methods in clinical practice for assessing a patient's cardiac and pulmonary functions, which involves measuring the distance that a patient can walk quickly on a flat and hard surface within 6 minutes.
The changes in the COPD assessment test (CAT) compared to the baseline. | 24 hours after administration, 4 and 12 weeks after the last administration.
  CAT is a self-completed questionnaire tool by the patients, used to assess the extent to which the condition of chronic obstructive pulmonary disease affects their quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No